CLINICAL TRIAL: NCT05031637
Title: Home Blood Pressure During Night-time Sleep as a Better Treatment Target for Patients With Hypertension: a Proof-of-concept Randomized Controlled Trial
Brief Title: Using Night-time Blood Pressure to Treat Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lee Kam Pui, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021.253-T
Record Dates: First submitted 2021-08-29; First posted 2021-09-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Hypertension
Keywords: hypertension; ABPM; nocturnal hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment by night-time BP (Experimental): titrate drug treatment in the evening against night home blood pressure monitoring (HBPM) SBP (aiming SBP of <120 mmHg; intervention group)
  Interventions: Behavioral: treatment of BP by using night-time BP
- treatment by daytime BP (Other): Usual care - titrate drug treatment in the morning against HBPM SBP (aiming SBP of <135 mmHg; control group)
  Interventions: Behavioral: treatment of BP by using daytime BP

INTERVENTIONS:
Behavioral: treatment of BP by using night-time BP — titration of BP medications to target according to night-time SBP
  Arms: treatment by night-time BP
Behavioral: treatment of BP by using daytime BP — titration of BP medications to target according to daytime SBP
  Arms: treatment by daytime BP

SUMMARY:
Objectives: To examine the feasibility of conducting night-time home blood pressure(BP) monitoring (during sleep) and titration of medications in the evening. This will provide data for sample size calculation for the main trial, which will examine whether night-time BP is a better target than conventional daytime BP for hypertension management.

Hypothesis to be tested: night-time home BP monitoring(HBPM) and evening drug titration are acceptable to patients; and future main trial is feasible in terms of recruitment/dropout rate/medication adherence.

Design and subjects: This pilot randomized-controlled trial will recruit 78 patients with nocturnal hypertension (asleep systolic BP 120mmHg on ambulatory blood pressure monitoring(ABPM)). They will be allocated in 1:1 ratio to have their medication titrated in the evening according to night HBPM (Experimental group) or in the morning according to daytime HBPM (control group) respectively.

Instruments: ABPM/HBPM. Interventions: titration of the dose(s) of anti-hypertensive medications in the evening according to night HBPM (experimental group) and in the morning according to daytime HBPM (control group) every 4 weeks.

Main outcome measures: ABPM at baseline and at 6 months Data analysis and expected results: The rate of recruitment/dropout and adherence to night HBPM will be presented. The feasibility of HBPM will be assessed by the patients' adherence to HBPM and by patients' interviews. ANCOVA will be used to evaluate whether titration of medication can normalize BP levels. We expect patients to have a high adherence rate and that titration of evening doses of medications will better improve night-time BP on ABPM.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed hypertension (HT) from clinical records
* nocturnal HT (night-time systolic blood pressure (SBP) during sleep ≥120 mmHg) and stage I hypertension (daytime SBP = 135-159mmHg)

Exclusion Criteria:

* patients with atrial fibrillation (many home blood pressure (BP) machines are not validated in these patients and these patients have greater BP variability)
* daytime office systolic BP ≥180 mmHg or diastolic BP ≥120 mmHg (regardless of nocturnal BP) because these patients need urgent BP treatment and it is not known if medications given in the evening are equally effective
* patients with known obstructive sleep apnoea because the night-time BP of these patients is predominately affected by the sleep apnoea
* patients with known stroke, ischemic heart disease, heart failure, kidney failure, peripheral vascular disease and diabetes mellitus because their daytime BP targets will be different
* dementia or psychiatric illness that impairs patients' ability to perform home blood pressure monitoring (HBPM) by themselves
* patients with end-stage malignancies
* nocturnal worker, because they will have a reverse BP pattern to other participants
* patients who sleep after 2am or wake up before 4am because these patients will not be asleep during night HBPM
* patients receiving ≥3 BP medications at maximal tolerated doses because there is little space for drug titration and these patients may have secondary HT representing another disease spectrum
* patients receiving anti-coagulants because ABPM can induce significant bruises (during repeated cuff inflations) in these patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
the rate of recruitment | 0 month to 18 month (anticipated recruitment period)
  number of participants recruited per month during recruitment period
feasibility of home blood pressure (BP) measurement | 0 month to 24 month (end of trial)
  the proportion of patients who can measure nocturnal BP successfully
feasibility of repeated ambulatory blood pressure monitoring (ABPM) | 0 month to 24 month (end of trial)
  the proportion of patients finished both ABPM
dropout rate | 0 month to 24 month (end of trial)
  number of participants drop-out from each arm

SECONDARY OUTCOMES:
systolic BP (SBP) / diastolic BP (DBP) on ABPM | taken at 0 month and 6 month for each patient
  Mean daytime/night-time/24-hour SBP/DBP
serum creatinine level | taken at 0 month and 6 month
  an assessment for renal function (the higher value suggest poorer renal function)
lipid profile | taken at 0 month and 6 month
  low-density lipoprotein (LDL), high-density lipoprotein (HDL), Triglyceride (TG), total cholesterol (TC)
microalbuminuria | taken at 0 month and 6 month
  the presence of microalbuminuria suggest renal damage

CONTACTS AND LOCATIONS:
Locations (1):
- School of public health and primary care, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
will share data on responsible requests